CLINICAL TRIAL: NCT02015897
Title: Effect of Physical Therapy on Breast Cancer Related Lymphedema; A Multicenter, Randomized, Single-blind, Equivalence Trial
Brief Title: Effect of Physical Therapy on Breast Cancer Related Lymphedema
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Esbjerg Hospital - University Hospital of Southern Denmark (Other)
Responsible Party: Principal Investigator, Valgerdur Hilmarsdottir Gram, Associate Professor, PhD, Esbjerg Hospital - University Hospital of Southern Denmark
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: S-20130091
Record Dates: First submitted 2013-12-03; First posted 2013-12-19 (Estimated); Last update posted 2023-01-31 (Actual); Status verified 2023-01

CONDITIONS: Lymphoedema; Breast Cancer
MeSH Terms: conditions — Lymphedema; Breast Neoplasms

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Physical TherapyB (Active Comparator): Group B
  Interventions: Procedure: Physical TherapyA
- Physical TherapyA (Placebo Comparator): Group A
  Interventions: Procedure: Physical TherapyB

INTERVENTIONS:
Procedure: Physical TherapyA — Group A:
  * Skin care
  * Manual lymphatic drainage
  * Bandaging using Coban™2Lite
  * Guidance on physical activity
  Arms: Physical TherapyB
Procedure: Physical TherapyB — Group B:
  * Skin care
  * Bandaging using Coban™2Lite
  * Guidance on physical activity
  Arms: Physical TherapyA

SUMMARY:
The objective of this study is to investigate if Complete Decongestive Therapy is equally effective whether it includes manual lymphatic drainage or not in the treatment of lymphoedema among patients with breast cancer.

DETAILED DESCRIPTION:
Physical therapy treatment of patients with lymphoedema includes treatment based on the principles of 'Complete Decongestive Therapy' (CDT). CDT consists of following components; skin care, manual lymphatic drainage, bandaging and exercises. Regarding what type of treatment of treatments is most effective, the scientific evidence is sparse. Studies have focused on the time-consuming manual lymphatic drainage, but the scientific evidence is not consistent.

A randomized, single-blind, equivalence trial. A total of 160 breast cancer patients with lymphoedema will be recruited from 3 hospitals and randomised into one of two treatment groups: A: Complete Decongestive TherapyA (incl. manual drainage) or B: Complete Decongestive TherapyB (except manual lymphatic drainage

ELIGIBILITY:
Inclusion Criteria:

* The diagnose breast cancer regardless of date for operation and identified lymphoedema
* Precede ultrasonic scanning of axilla in order to exclude local relapse
* Lymphoedema > 2 cm i.e. stage II-III
* Completed radiotherapy and/or chemotherapy at least 2 months prior inclusion

Exclusion Criteria:

* Relapse of breast cancer
* Untreated infection
* Untreated heart failure
* Untreated renal failure
* Untreated deep venous thrombosis in the arm
* Unable to participate in physiotherapy treatment and/or not able to understand instructions

Ages: 18 Years to 90 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2014-01; Primary Completion 2017-09-01 (Actual); Study Completion 2017-09-01 (Actual)

PRIMARY OUTCOMES:
The percentage volume reduction of lymphoedema (%) | 7 months

SECONDARY OUTCOMES:
Differences in circumference of the arm (composite outcome measure), bodyweight, patient sensation of heaviness, patient sensation of tension, and quality of life | 7 months
  Circumference of the arm consists of 7 measurements but these will be converted to one outcome measure when estimating the difference between baseline and post intervention measurements

OTHER OUTCOMES:
Percentage volume reduction of lymphedema (%) from baseline to week 4. Percentage volume reduction of lymphedema (%) from week 4 to week 7 | 7 months

CONTACTS AND LOCATIONS:
Overall Officials: Bibi Gram, PhD, Study Director — THe Hospital of Southwest Denmark
Locations (3):
- Denmark (3):
  - Hospital of Southwest Denmark, Esbjerg, Region Syddanmark
  - Department of Rehabilitation, Odense University Hospital, Odense, Region Syddanmark
  - Department of Physical Therapy, Lillebaelt Hospital, Vejle, Region Syddanmark

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Tambour M, Holt M, Speyer A, Christensen R, Gram B. Manual lymphatic drainage adds no further volume reduction to Complete Decongestive Therapy on breast cancer-related lymphoedema: a multicentre, randomised, single-blind trial. Br J Cancer. 2018 Nov;119(10):1215-1222. doi: 10.1038/s41416-018-0306-4. Epub 2018 Oct 24. PMID 30353049
- [Derived] Tambour M, Tange B, Christensen R, Gram B. Effect of physical therapy on breast cancer related lymphedema: protocol for a multicenter, randomized, single-blind, equivalence trial. BMC Cancer. 2014 Apr 3;14:239. doi: 10.1186/1471-2407-14-239. PMID 24708851
- See also: Link to the Hospital of Southwest Denmark — http://www.sydvestjysksygehus.dk